CLINICAL TRIAL: NCT03369496
Title: The Montreal Neighbourhood Networks and Healthy Aging Panel (MoNNET-HA)
Brief Title: The Montreal Neighbourhood Networks and Healthy Aging Panel
Acronym: MoNNET-HA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Spencer Moore, Associate Professor, Queen's University
Other Study IDs: GPHE-148-13; MOP-84584 (Other Grant/Funding Number: Canadian Institutes of Health Research); CHL-126208 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2017-12-01; First posted 2017-12-12 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Obesity; Depression; Physical Activity; Hypertension; Health Behavior; Subjective Health
Keywords: Social Capital; Social Support; Neighborhood; Population Health; Healthy Aging; Adult; Canada
MeSH Terms: conditions — Obesity; Depression; Motor Activity; Hypertension; Health Behavior | interventions — Neighborhood Characteristics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MoNNET-HA Panel: Adults 25 years and older residing in the Montreal Metropolitan Area
  Interventions: Other: Social capital; Neighborhood environment

INTERVENTIONS:
Other: Social capital; Neighborhood environment — Observational study examining the relationship among neighborhood environment, social capital and health among Montreal adults

SUMMARY:
Social networks, social capital, i.e., network-accessed resources, and neighbourhood environments have been shown associated with a range of health behaviours and conditions, including obesity, physical activity, nutrition, and mental health. Research on social capital and health in Montreal has shown the importance of network social capital for a person's subjective health status, sense of control, self-reported physical activity, and obesity. Research has also shown high social capital to reduce health service use, mental health service use, and improve the management of chronic illnesses. Despite advances in the understanding of social capital and its link to health and health service use, most research on social capital is cross sectional and is unable to identify the causal pathways linking social networks and capital to health and health care use. Longitudinal research would strengthen the evidence base for designing interventions to prevent or delay the use of health services, particularly in older adults.

This research has three main objectives: (1) transform the original sample of Montreal Neighbourhood Networks and Healthy Aging (MoNNET-HA) households (n=2707) into a panel study, (2) link the MoNNET-HA participant data to their Quebec Health Insurance Registry (Régie de l'assurance maladie (RAMQ)) information, and (3) assess the feasibility of extending the MoNNET-HA panel by one wave to include participant's core network members. Unique about the original MoNNET-HA sample is that it purposefully oversampled older adults (> 64 years old) but remains representative of Montreal adults at various ages and income levels. In addition, MoNNET-HA data is integrated into a GIS database which allows researchers to examine the effects of neighbourhood environmental characteristics on health. By linking MoNNET-HA data to RAMQ, researchers will be able to examine patterns of diagnosed health conditions, (e.g., fractures, depression), pharmaceutical use and adherence, and formal health care use over time. Transforming the cross-sectional study into a panel study would also allow researchers to examine longitudinally the dynamics of health and health care utilization among Panel participants over the life course, and the causal pathways linking neighbourhoods and networks to health and health care use.

ELIGIBILITY:
Inclusion Criteria:

* Adults 25 years and older,
* Residents of the Montreal Metropolitan Area, Canada,
* Had to reside at current residence for at least one year

Exclusion Criteria:

* Non- French or English-speaking households
* Institutionalized

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population-based sample of adults randomly selected using a 2-stage stratified cluster sampling strategy.
  1. In the first stage, 862 Montreal Metropolitan Area census tracts were stratified using the census-tract median income into tertile of high, medium and low income census tract areas. From each tertile, 100 census tracts were selected at random from each census-tract group for a total of 300 tracts.
  2. Within each selected census tract, three respondents were selected at random using from the 25-44 years age category, three respondents from the 45-64 years age category, and three respondents from the age group 65 years and older. This resulted in a total of 9 respondents per census tract and a total of 2707 respondents the MoNNET Panel.
Sampling Method: Probability Sample
Enrollment: 2707 (Actual)
Dates: Start 2007-07-01 (Actual); Primary Completion 2008-08-15 (Actual); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Obesity | Change from wave one obesity at wave two (2010) and wave three (2013)
  Self-reported height and weight converted to BMI with obesity =>30
Change in Depression | Change from wave one depression at wave two (2010) and wave three (2013)
  Center for Epidemiological Studies Depression 10-item Binary Scale; Depression was =>4
Change in Physical inactivity | Change from wave one physical inactivity at wave two (2010) and wave three (2013)
  International Physical Activity Questionnaire (IPAQ) was used to measure a person's metabolic equivalent of task (MET) over a one-week period; Physical inactivity was defined as having a MET of less than 600.
Change in Hypertension | Change from wave one hypertension at wave two (2010) and wave three (2013)
  Self-reported doctor-diagnosed hypertension
Change in Subjective Health | Change from wave one subjective health at wave two (2010) and wave three (2013)
  Self-reported health: 5 response options: Excellent, Very Good, Good, Fair, Poor

CONTACTS AND LOCATIONS:
Overall Officials: Spencer Moore, PhD, Principal Investigator — Queen's University (at time of study)

IPD SHARING:
Plan to Share IPD: Undecided
Discussions currently taking place.

REFERENCES:
- [Result] Moore S, Bockenholt U, Daniel M, Frohlich K, Kestens Y, Richard L. Social capital and core network ties: a validation study of individual-level social capital measures and their association with extra- and intra-neighborhood ties, and self-rated health. Health Place. 2011 Mar;17(2):536-44. doi: 10.1016/j.healthplace.2010.12.010. Epub 2010 Dec 16. PMID 21208822
- [Result] Leroux JS, Moore S, Richard L, Gauvin L. Physical inactivity mediates the association between the perceived exercising behavior of social network members and obesity: a cross-sectional study. PLoS One. 2012;7(10):e46558. doi: 10.1371/journal.pone.0046558. Epub 2012 Oct 2. PMID 23056343
- [Result] Legh-Jones H, Moore S. Network social capital, social participation, and physical inactivity in an urban adult population. Soc Sci Med. 2012 May;74(9):1362-7. doi: 10.1016/j.socscimed.2012.01.005. Epub 2012 Feb 22. PMID 22410270
- [Result] Bassett E, Moore S. Gender differences in the social pathways linking neighborhood disadvantage to depressive symptoms in adults. PLoS One. 2013 Oct 17;8(10):e76554. doi: 10.1371/journal.pone.0076554. eCollection 2013. PMID 24146888
- [Result] Bassett E, Moore S. Social capital and depressive symptoms: the association of psychosocial and network dimensions of social capital with depressive symptoms in Montreal, Canada. Soc Sci Med. 2013 Jun;86:96-102. doi: 10.1016/j.socscimed.2013.03.005. Epub 2013 Mar 19. PMID 23608098
- [Result] Moore S, Stewart S, Teixeira A. Decomposing social capital inequalities in health. J Epidemiol Community Health. 2014 Mar;68(3):233-8. doi: 10.1136/jech-2013-202996. Epub 2013 Nov 20. PMID 24258198
- [Result] Bassett E, Moore S. Neighbourhood disadvantage, network capital and restless sleep: is the association moderated by gender in urban-dwelling adults? Soc Sci Med. 2014 May;108:185-93. doi: 10.1016/j.socscimed.2014.02.029. Epub 2014 Feb 19. PMID 24650740
- [Result] Moore S, Teixeira A, Stewart S. Effect of network social capital on the chances of smoking relapse: a two-year follow-up study of urban-dwelling adults. Am J Public Health. 2014 Dec;104(12):e72-6. doi: 10.2105/AJPH.2014.302239. Epub 2014 Oct 16. PMID 25320891
- [Result] Moore S, Buckeridge DL, Dube L. Cohort Profile: The Montreal Neighbourhood Networks and Healthy Aging (MoNNET-HA) study. Int J Epidemiol. 2016 Feb;45(1):45-53. doi: 10.1093/ije/dyu137. Epub 2014 Jul 1. PMID 24984955
- [Result] Child S, Stewart S, Moore S. Perceived control moderates the relationship between social capital and binge drinking: longitudinal findings from the Montreal Neighborhood Networks and Health Aging (MoNNET-HA) panel. Ann Epidemiol. 2017 Feb;27(2):128-134. doi: 10.1016/j.annepidem.2016.11.010. Epub 2016 Dec 9. PMID 28027881